CLINICAL TRIAL: NCT03496181
Title: Graph Theoretical Analysis of Pre-operative fMRI Data in Bilingual Patients With Brain Tumors
Brief Title: Evaluation of Functional Magnetic Resonance Imaging (fMRI) in Patients Who Speak Two Languages Fluently
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-121
Record Dates: First submitted 2018-04-03; First posted 2018-04-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Glioma; Glioma of Brain; Glioma of Spinal Cord
Keywords: fMRI; MRI; 18-121; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Glioma | interventions — Language Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bilingual Participants with Glioma: Bilingual (English and Spanish speaking) patients will be recruited from the clinical service of the Department of Neurosurgery of MSK. All patients on the Neurosurgery service scheduled to undergo a resection of a tumor in or adjacent to the primary language areas will be screened to participate in this study.
  The study will be performed in concert with patient's regularly scheduled clinical care for his/her brain tumor. Clinical care (which will be performed whether or not the patient participates in the current study) will include: 1) pre-operative routine (anatomical) MRI and fMRI, 2) the surgery to remove the tumor, 3) intra-operative cortical stimulation to identify the essential motor and/or language areas. It should be stressed that neither the brain tumor surgery, nor the intra-operative cortical mapping will be changed in any way from routine practice.
  Interventions: Behavioral: Multilingual Aphasia Examination; Diagnostic Test: Language paradigms + RS fMRI
- Healthy Volunteers: Normal, healthy volunteers who express interest in participation and who meet the eligibility criteria will be recruited for this study. It is anticipated that healthy volunteers will mostly consist of medical professionals. They will consist of 10 monolinguals (defined as native English speakers), 10 early bilinguals (defined as acquiring proficiency in the second language before 10 years of age), and 10 late bilinguals (defined as acquiring proficiency in the second language after 10 years of age).
  Interventions: Diagnostic Test: Language paradigms + RS fMRI + one anatomical sequence

INTERVENTIONS:
Behavioral: Multilingual Aphasia Examination — For patients only prior to MRI scans.
  The MAE contains eleven subtests in five categories which may be used to assess both languages in bilinguals and the participant's primary language in monolinguals: Oral Expression, Spelling, Oral Verbal Understanding, Reading, and Rating Scales. Subtests are scored for accuracy of individual items on a three-point scoring system (0, 1, 2). Contained within these domains are The Token Test, Aural Comprehension of Words and Phrases and Visual Naming which naturally parallel fMRI and direct cortical stimulation behavioral assays already in place for clinical use (phonemic fluency, auditory responsive naming and confrontation naming respectively). The MAE is expected to take under 50 minutes.
  Groups: Bilingual Participants with Glioma
Diagnostic Test: Language paradigms + RS fMRI — 10 monolingual patients: 2 language paradigms + RS fMRI = 7x3 = 21 minutes 10 early bilingual patients: 2 language paradigms+ RS fMRI = 7x3 = 21 minutes 10 late bilingual patients: 2 language paradigms+ RS fMRI = 7x3 = 21 minutes
  Groups: Bilingual Participants with Glioma
Diagnostic Test: Language paradigms + RS fMRI + one anatomical sequence — 10 monolingual English volunteers: 2 task language paradigms* + 1 Resting State fMRI + one anatomical sequence for a total of approximately 25 minutes.
  10 late bilingual volunteers: 4 language paradigms (2 English + 2 Spanish) + 1 Resting State fMRI + one anatomical sequence for a total of approximately 39 minutes.
  10 early bilingual volunteers: 4 language paradigms (2 English + 2 Spanish) + 1 Resting State fMRI + one anatomical sequence for a total of approximately 39 minutes.
  Groups: Healthy Volunteers

SUMMARY:
Functional magnetic resonance imaging (fMRI) is a non-invasive test used to detect changes in brain activity by taking picture of changes in blood flow. The imaging helps doctors better understand how the brain works. Task based fMRI (TB fMRI) prompts patients to perform different activities (e.g. word selection in a reading task), and is routinely performed on patients in preparation for a Neurological surgery (surgery that involves the nervous system, brain and/or spinal cord). The purpose is to locate areas of the brain that control speech and movement; these images will help make decisions about patient surgeries. However, there are however gaps in knowledge specific to the language areas of the brain, especially for non-English patients and bilingual patients (those who are fluent in more than one language). This study proposes to evaluate if resting state fMRI (RS fMRI) that does not require any tasks, along with a novel way to analyze these images using "graphy theory," may provide more information. Graph theory is a new mathematical method to analyze the fMRI data. The overall goal is to determine if graph theory analysis on RS fMRI may reduce differences in health care treatment and outcomes for non-English speaking and bilingual patients. We hope that the results of this study will allow doctors to perform pre-operative fMRI in patients who do not speak English.

ELIGIBILITY:
Inclusion Criteria:

All patients and volunteers will be recruited by listed consenting professionals. Volunteers do not need to be MSK employees.

* Patients/ healthy volunteers ≥ 18 years old
* Patients/ healthy volunteers must be able to perform the language paradigms on cue while inside the scanner
* Patients/ healthy volunteers who are monolingual English speakers, early bilinguals (English and Spanish) or late bilinguals (English and Spanish)
* Patients must be newly diagnosed with a glioma (from prior histology) or must be suspected to have a glioma on imaging (to be confirmed by post-operative histology)
* Patient's location of the tumor must involve the expected location of Broca's area (left pars opercularis and/or pars triangularis). This determination will be made on the basis of a pre-operative MRI by a fellowship-trained Neuroradiologist

Early bilingual will be defined as acquiring proficiency in the second language before 10 years of age.

Exclusion Criteria:

* Patients/ volunteers who are unable to comply or complete MRI exams as per the Department of Radiology's standard guidelines (e.g.: claustrophobia, high levels of anxiety, pacemaker etc.)
* Patient/ volunteers who are unable to perform the language paradigms on cue while inside the scanner (due to weakness, deafness, inability to understand or follow instructions etc.)
* Volunteers with a history of neurological disorders, psychiatric disorders or cancer
* Female patients/ volunteers who are pregnant or nursing
* Patients/ volunteers from the vulnerable population, as defined by 45 CFR 46

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research participants will be identified by a member of the patient's treatment team, listed protocol investigators, or Neuroradiology research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Comparison of RS fMRI and overall TB fMRI | Through study completion, an average of 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Holodny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - City College of New York, New York, New York
- IMT School of Advance Studies Lucca, Lucca, Lucca LU, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03496181/ICF_000.pdf